CLINICAL TRIAL: NCT06758128
Title: Role of Immunity and Genetic Predisposition in Chronic Heart Failure Exacerbation
Brief Title: Genetic and Immunity in Heart Failure
Acronym: GISCO
Status: Recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 6721
Record Dates: First submitted 2024-12-24; First posted 2025-01-03 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2024-12

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Genetic: Evaluation of HS1,2 polymorphisms — Echocardiograms will be performed by experienced operators of the echocardiography service.
  Inflammatory profile. A single additional blood sample (3 cc) will be collected. Plasma will be isolated from whole blood to determine pro-inflammatory cytokines.
  Immunoprofile: Circulating lymphocytes will be separated according to Ficoll gradient (into the two different components of immunity (B and T lymphocytes) with different inflammatory phenotypes.
  Evaluation of HS1,2 polymorphisms and estrogen levels: DNA purifications and amplifications will be performed from an aliquot of the single whole blood sample. Genomic DNA will be isolated using the QIAamp DNA Mini and Blood Mini kit (QIAGEN Hilden, Germany) according to the manufacturer's protocol. 9 single nucleotide polymorphisms (SNPs) in four specific polymorphic regions of the 3'-1 Regulatory Region (3'RR-1) of the human immunoglobulin (IgH) heavy chain locus will be sequenced.
  Other Names: Cytofluorimetric immunoprofile; Echocardiography

SUMMARY:
Heart failure is a major health problem with serious consequences on mortality and morbidity worldwide. In chronic heart failure an alteration of the inflammatory state occur. The aim of this study will be to describe the relationship between markers of inflammation in patients with heart failure with preserved ejection fraction, gender differences and advanced age.

The study sample will include patients hospitalized in the Unit of General Medicine and Aging with a diagnosis of heart failure based on the guidelines. Clinical and demographic data will be collected from the electronic records of our hospital system. A complete history will be obtained, including the possible etiology of heart failure, cardiac and noncardiac comorbidities, all medications, intracardiac devices, and chronic oxygen treatment. All patients will be documented for peripheral edema, pulmonary rales and jugular vein distension. NYHA (New York Heart Association) class will be identified at discharge. In addition, a blood sample will be taken to obtain a complete panel including total blood count, glycemia, renal function, electrolytes and liver function tests, as per standardized clinical practice. NT-proBNP (Amino-terminal pro Natriuretic Peptide B) will be measured at admission and discharge from the hospital, as per standardized clinical practice.

Echocardiograms will be performed by experienced operators of the echocardiography service of our Polyclinic, according to the American Society of Echocardiography guidelines.

A single additional blood sample will be collected during one of the normal routine blood draws for all immunological tests. Plasma from each participant will be isolated to determine the concentrations of several cytokines. Circulating lymphocytes will be separated according to Ficoll gradient (peripheral blood mononuclear cells, PBMC) into the two different components of immunity (B and T lymphocytes) with different inflammatory phenotypes Evaluation of enhancer (HS)1,2 polymorphisms and estrogen levels: DNA purifications and amplifications will be performed from an aliquot of the single whole blood sample collected for the evaluation of the inflammatory profile. Genomic DNA will be isolated and 9 SNPs in four specific polymorphic regions of the 3'-1 Regulatory Region (3'RR-1) of the human immunoglobulin (IgH) heavy chain locus will be sequenced. Follow-up will be performed by telephone contacting the patients or their caregivers 90 days after discharge.

ELIGIBILITY:
Inclusion criteria:

* Adult patients (age ≥18 years) with exacerbation of chronic heart failure with reduced or preserved ejection fraction,
* stable haemodynamic conditions, without the need for inotropic support at the time of admission to the ward,
* signature of the informed consent.

Exclusion criteria:

. age <18 years;

* pregnancy;
* acute coronary syndromes;
* end-stage renal failure (clearance <30 mL/min) or dialysis;
* ongoing sepsis;
* bed rest syndrome;
* any concomitant neoplasm,
* congenital and acquired immunodeficiencies (HIV, immunosuppressive drugs).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study sample will include adult patients (>18 years) hospitalized in the Unit of General Medicine and Aging with a diagnosis of heart failure based on the guidelines on heart failure. Clinical and demographic data will be collected from the electronic records of our hospital information system. The medical record of each patient will be used to record demographic and clinical characteristics, data relating to the presentation in the Emergency Department, the evaluation and any event that occurred during hospitalization, including the conditions at discharge.
Sampling Method: Probability Sample
Enrollment: 215 (Estimated)
Dates: Start 2025-02-04 (Actual); Primary Completion 2026-07-15 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Prevalence of HS1,2 enhancer alleles of human immunoglobulin heavy chains in patients with heart failure | 6 months
  Difference in the prevalence of HS1,2 enhancer alleles of human immunoglobulin heavy chains in patients with heart failure with preserved ejection fraction and in patients with heart failure with reduced ejection fraction.
Inflammatory markers in heart failure | 6 months
  To evaluate any differences in inflammatory markers in patients with heart failure with preserved ejection fraction and reduced ejection fraction, with particular attention to gender and age differences.

SECONDARY OUTCOMES:
Genetic polymorphisms and estrogen levels | 6 months
  Evaluate the association between different genetic polymorphisms and estrogen levels in different models of patients with chronic heart failure with preserved and reduced ejection fraction

CONTACTS AND LOCATIONS:
Overall Officials: Rossella Cianci, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS
Locations (2):
- Italy (2):
  - IRCCS Casa Sollievo della Sofferenza, San Giovanni Rotondo, Foggia
  - Fondazione Policlinico Universitario A. Gemelli IRCCS, UOC Medicina Genarale e dell'Invecchiamento, Rome, Lazio